CLINICAL TRIAL: NCT05039918
Title: The Healing Power of Touch: Investigation of a Peripheral Neurological Mechanism for Reducing Pain and Enhancing Neurodevelopmental Outcomes
Brief Title: Neonatal Experience of Social Touch
Acronym: NEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool Women's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 21LJMUSPONSOR051; 291417 (Other: IRAS)
Record Dates: First submitted 2021-08-03; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Premature Birth; Infant Development; Pain
Keywords: CT Fibres; Affective touch
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Allocation sequence will be randomised in advance by a trusted member of LJMU staff who is not involved in the study, using a computerised website to generate random numbers. The sequences will be placed in sealed opaque envelopes and stored in a secure location on-site. The use of an off-site computerised system for group allocation will decrease the risk of allocation bias. Eligible infants whose person(s) with parental responsibility have provided consent will be assigned the next available envelope which will be accessed by the lead researcher prior to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Following randomisation, infants will receive CT-optimal stimulation (gentle stroking) at a velocity of 3cm/s over the area which the infant will be stroked (10cm) for a duration of 10s applied proximally to the pain site prior to the heel prick. Location of the heel prick will be based on clinical judgement. There will be an inter-stimulus interval of approximately 1 second between the end of the touch and heel prick, and touch stimulation will be applied to the lower leg ipsilateral to the heel receiving the noxious stimuli. All infants will have cardio-respiratory monitoring during the intervention. All other environmental factors will be as standard care (e.g., temperature, lighting and sounds).
  The heel prick will be performed by a member of the infants designated clinical team who have performed the procedures in a standardised manner according to the institutional and unit policy.
  Interventions: Behavioral: Affective touch
- Control (No Intervention): Infants who are randomised to the control group will receive standard care consistent with neonatal policy. The infant will undergo a heel prick in the incubator or crib in an identical fashion to the infants in the intervention group.

INTERVENTIONS:
Behavioral: Affective touch — Gentle stroking at CT-optimal speed
  Arms: Intervention

SUMMARY:
The purpose of this randomised control trial is to determine the efficacy of CT-optimal touch (gentle stroking at 3cm/s) for newborn's who require a heel prick.

DETAILED DESCRIPTION:
Newborn infants are subject to several novel experiences that cause physiological, biochemical and behavioural indicators of stress; even routine and common events such as handling, changing a diaper or being bathed can increase salivary cortisol levels. Excluding surgery and mechanical ventilation, the most common procedural pain sources in newborns are heel-lancing and venepuncture. Tactile interventions such as skin to skin care and 'still containment hold' are widely used in clinical care with apparent positive results such as lower mean respiratory heart rate and pain measures, and higher oxygen saturation; yet, dynamic touch interventions have reported to be more beneficial than static touch interventions.

A distinct type of nerve fibres, CT (C tactile) afferents, found exclusively in hairy skin, that respond optimally to gentle stroking at a velocity of ~1-10cm/s, are part of a system for processing pleasant and social rewarding touch. CT fibre activation also plays a role in pain inhibition and may be linked to the development of self-regulation, thereby, serving a neuroprotective function for the developing infant brain. Here we will investigate whether tactile stimulation at CT-optimal velocity will reduce biochemical and physiological indicators of stress in infants, as determined by salivary cortisol, heart rate and blood oxygenation levels.

ELIGIBILITY:
Inclusion Criteria:

* The infant is born between 35 and 42 weeks.
* Require a heel prick
* Infants may be treated with antibiotics.
* Infants may be supported with non-invasive respiratory support.
* Infants may require blood sugar monitoring.
* Infants may be monitored for jaundice or infection.
* Written consent has been obtained from the person(s) with parental responsibility.

Exclusion Criteria:

* Have a history of neurological problems.
* Receiving pharmacological analgesics.
* Known genetic condition.
* Breastfed babies
* Admitted to high dependency or intensive care
* Invasive respiratory support
* Receiving parenteral nutrition
* Has received any treatment for seizures
* Clinical instability in the judgment of nurses/midwives and paediatricians looking after the baby and mother.

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Salivary cortisol | Immediately before heel prick and 20 minutes after
  Change between cortisol levels at baseline and 20 minutes after

SECONDARY OUTCOMES:
Heart rate | Baseline, time of event, 20 mins after and 60 minutes after
  Change from baseline heart rate to to time of event and two post test periods
Blood oxygenation | Baseline, time of event, 20 mins after and 60 minutes after
  Change from baseline oxygenation levels to time of event and two post test periods

CONTACTS AND LOCATIONS:
Overall Officials: Francis McGlone, Professor, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool Women's Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manzotti A, Cerritelli F, Esteves JE, Lista G, Lombardi E, La Rocca S, Gallace A, McGlone FP, Walker SC. Dynamic touch reduces physiological arousal in preterm infants: A role for c-tactile afferents? Dev Cogn Neurosci. 2019 Oct;39:100703. doi: 10.1016/j.dcn.2019.100703. Epub 2019 Aug 21. PMID 31487608
- [Background] Gursul D, Goksan S, Hartley C, Mellado GS, Moultrie F, Hoskin A, Adams E, Hathway G, Walker S, McGlone F, Slater R. Stroking modulates noxious-evoked brain activity in human infants. Curr Biol. 2018 Dec 17;28(24):R1380-R1381. doi: 10.1016/j.cub.2018.11.014. PMID 30562526